CLINICAL TRIAL: NCT03231397
Title: Noninvasive Assessment of Abdominal Aortic Aneurysm (AAA) Wall Structural Integrity and Inflammation as Predictors of Expansion and/or Rupture
Brief Title: Predictors of AAA Expansion and/or Rupture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We were unable to recruit more subjects who met the inclusion/exclusion criteria and we have closed the study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 201702141
Record Dates: First submitted 2017-06-22; First posted 2017-07-27 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: Abdominal Aortic Aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Eligible subjects in this study will have either a known abdominal aortic aneurysm (AAA) or because they do not have an AAA (control group).
  The purpose of this research study is to further study, through FEA, changes that occur in the mechanical properties of the aortic wall. The investigator will compare two radiotracers, 18F-FDG and 11C-PBR28 to determine if one provides more useful and reliable information about inflammation. 18F-FDG and 11C-PBR28 are radioactive drugs that will be used for imaging during the PET-CT scan. The investigator will also compare the results describing the mechanical properties of the AAA wall to the degree of inflammation in that wall as determined by PET-CT imaging to define new and better predictors of AAA growth and/or rupture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (Other): Six control subjects (three males and three females) with known atherosclerosis by standard clinical criteria without aneurysmal disease.
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Interventions: Drug: Assess AAA rupture risk by PET-CTA scans; Drug: 18F-fludeoxyglucose (FDG); Diagnostic Test: 11C-PBR28
- Small AAA's (Other): Six subjects (three males and three females) with small AAAs (diameter 3.0-4.5cm).
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Interventions: Drug: Assess AAA rupture risk by PET-CTA scans; Drug: 18F-fludeoxyglucose (FDG); Diagnostic Test: 11C-PBR28
- Rapidly expanding AAA's (Other): Six subjects (three males and three females) with rapidly expanding AAAs (>0.5cm over 6 months and/or >1.0cm over 12 months).
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Interventions: Drug: Assess AAA rupture risk by PET-CTA scans; Drug: 18F-fludeoxyglucose (FDG); Diagnostic Test: 11C-PBR28
- AAA's undergoing treatment (Other): Six subjects (three males, AAA >5.5cm and three females, AAA >5.0cm) with AAAs that are indicated for treatment.
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Interventions: Drug: Assess AAA rupture risk by PET-CTA scans; Drug: 18F-fludeoxyglucose (FDG); Diagnostic Test: 11C-PBR28

INTERVENTIONS:
Drug: Assess AAA rupture risk by PET-CTA scans — Assess AAA rupture risk by PET-CTA scans
Drug: 18F-fludeoxyglucose (FDG) — Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
  Other Names: 18F-FDG
Diagnostic Test: 11C-PBR28 — Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging

SUMMARY:
Eligible subjects in this study will have either a known abdominal aortic aneurysm (AAA) or because they do not have an AAA (control group).

The purpose of this research study is to further study, through FEA, changes that occur in the mechanical properties of the aortic wall. The investigator will compare two radiotracers, 18F-FDG and 11C-PBR28 to determine if one provides more useful and reliable information about inflammation. 18F-FDG and 11C-PBR28 are radioactive drugs that will be used for imaging during the PET-CT scan. The investigator will also compare the results describing the mechanical properties of the AAA wall to the degree of inflammation in that wall as determined by PET-CT imaging to define new and better predictors of AAA growth and/or rupture.

DETAILED DESCRIPTION:
Eligible subjects in this study will have either a known abdominal aortic aneurysm (AAA) or because they do not have an AAA (control group).

The aorta serves as the main artery to supply blood flow to the body. It is approximately the size of a garden hose. Due to the effects of high blood pressure (hypertension), atherosclerosis (hardening of the arteries), and tobacco use, the aorta may widen and enlarge to form an aneurysm. An abdominal aortic aneurysm (AAA) is a dilation (enlargement) or ballooning out of a section of blood vessel caused by disease or weakness in the wall of the aorta below the level of the kidney arteries. As an AAA dilates and increases in size, rupture of the AAA may occur. AAA rupture carries a significant risk of death.

Currently, aortic size is the primary factor used to assess aortic rupture risk. There are other imaging procedures (imaging modalities) that are being used and developed to assess AAA rupture risk. Finite element analysis (FEA) is a way to study the mechanical properties of the aortic wall, including areas of stress and strength that are used to calculate rupture risk. Positron Emission Tomography (PET) utilizes glucose (a form of sugar) labeled with a radioactivity to look at the metabolic activity and inflammation in the aortic wall.

The purpose of this research study is to further study, through FEA, changes that occur in the mechanical properties of the aortic wall. The investigator will compare two radiotracers, 18F-FDG and 11C-PBR28 to determine if one provides more useful and reliable information about inflammation. 18F-FDG and 11C-PBR28 are radioactive drugs that will be used for imaging during the PET-CT scan. The investigator will also compare the results describing the mechanical properties of the AAA wall to the degree of inflammation in that wall as determined by PET-CT imaging to define new and better predictors of AAA growth and/or rupture.

The radioactive tracers that are used in this study are 18F-fludeoxyglucose (FDG) and 11C-PBR28 (PBR) which stands for Peripheral Benzodiazepine Receptor. 11C-PBR28 is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration. FDG is an approved drug by the FDA, however in this study it is considered investigational.

Goal: Twenty-four subjects will be recruited for this study. Six control subjects (three males and three females), will be considered. Control subjects will have known atherosclerosis, without aneurysmal disease. Six subjects (three males and three females) with small AAAs (diameter 3.0-4.5cm), six subjects (three males, AAA >5.5cm and three females, AAA >5.0cm) with AAAs that are indicated for treatment, and six subjects (three males and three females) with rapidly expanding AAAs (>0.5cm over 6 months and/or >1.0cm over 12 months) will be considered.

Subjects will have blood drawn to perform a genetic test that will look at genes and proteins to determine subject eligibility. Once the blood work is assessed for eligibility, subjects will undergo the PET-CT scan. The imaging will take approximately 3 hours to complete.

ELIGIBILITY:
Inclusion

* All ethnic groups
* 45 years of age or older
* *Must fit into one of the three following groups:

  * Control group (atherosclerosis without aneurysmal disease
  * Small AAA (3-4.5 cm)
  * Rapidly growing AAA (0.5 cm in 6 months or 1 cm in 12 months)

Exclusion

* At risk population (cognitively impaired)
* Any exclusion for PT-CT (i.e., allergy to contrast)
* Any woman planning to become pregnant, suspects pregnancy, pregnant or breastfeeding)
* Any greater than normal potential for cardiac arrest
* Renal disease (eGFR <60 mg/ml/1.73m2)
* Claustrophobic reactions and/or is unable to lie on the exam table for 60 minutes
* Significant radiation exposure via other trials or medical testing

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean J. English, MD, Principal Investigator — Washington University School of Medicine, St. Louis, MO 63110
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The plan was to enroll 30 subjects, however, due to the lack of willing participants, we were only able to enroll 2 subjects.
Groups:
- Control Group: Six control subjects (three males and three females) with known atherosclerosis by standard clinical criteria without aneurysmal disease.
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Assess AAA rupture risk by PET-CTA scans: Assess AAA rupture risk by PET-CTA scans
  18F-fludeoxyglucose (FDG): Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
  11C-PBR28: Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
- Small AAA's: Six subjects (three males and three females) with small AAAs (diameter 3.0-4.5cm).
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Assess AAA rupture risk by PET-CTA scans: Assess AAA rupture risk by PET-CTA scans
  18F-fludeoxyglucose (FDG): Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
  11C-PBR28: Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
- Rapidly Expanding AAA's: Six subjects (three males and three females) with rapidly expanding AAAs (>0.5cm over 6 months and/or >1.0cm over 12 months).
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Assess AAA rupture risk by PET-CTA scans: Assess AAA rupture risk by PET-CTA scans
  18F-fludeoxyglucose (FDG): Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
  11C-PBR28: Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
- AAA's Undergoing Treatment: Six subjects (three males, AAA >5.5cm and three females, AAA >5.0cm) with AAAs that are indicated for treatment.
  To assess AAA rupture risk by PET-CTA scans, participants will undergo PET-CT scan using 11C-PBR28 and 18F-fludeoxyglucose (FDG) tracer. Participants will have a blood draw for genetic testing, pregnancy testing if female and creatinine testing.
  Assess AAA rupture risk by PET-CTA scans: Assess AAA rupture risk by PET-CTA scans
  18F-fludeoxyglucose (FDG): Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
  11C-PBR28: Assess AAA rupture risk by PET-CTA scans using 18F-fludeoxyglucose (FDG)and 11C-PBR28 PET-CT and contrast-enhanced CTA imaging
Period: Overall Study
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment
Started | 0 | 1 | 1 | 0
Completed | 0 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to enroll subjects in the control group and the AAA's undergoing treatment who met the inclusion/exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment | Total
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 |  | 0
  Between 18 and 65 years |  | 0 | 0 |  | 0
  >=65 years |  | 1 | 1 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 |  | 0
  Male |  | 1 | 1 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 |  | 0
  Asian |  | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 |  | 0
  Black or African American |  | 0 | 0 |  | 0
  White |  | 1 | 1 |  | 2
  More than one race |  | 0 | 0 |  | 0
  Unknown or Not Reported |  | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Standard Uptake Value (SUV)
Description: Aortic inflammation as demonstrated by uptake of radiotracer
Time Frame: 1 day
Population: Recruitment was difficult. We enrolled 1 subject with a small AAA and 1 subject with a rapidly expanding AAA, however, we were unable to recruit the number of subjects in each category to provide meaningful outcomes.
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Rupture Potential Index (RPI)
Description: Rupture potential index (RPI) is defined as the ratio of the acting wall stress to the wall strength, and the maximum RPI for AAA represents its rupture risk. Currently, the primary factor considered for risk of human AAA rupture is aortic diameter; however, it is well documented that small AAAs (<5cm) rupture, while many large AAAs (>8cm) are incidentally discovered.
  We will assess the ability of imaging techniques to determine abdominal aortic aneurysm (AAA) rupture risk individually and in concert.
Time Frame: 9-10 months
Population: as for outcome 1
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Qualitative Comparison of SUV and RPI
Description: Finite element analysis (FEA) is a computerized numerical method used for the prediction of how the aorta may behave under stress. This software will be used to assess the same aortic volume comparing areas of greatest stress and lowest strength. Co-registration of images obtained by different imaging modalities will allow for comparison between imaging modalities. With direct co-registration of the data sets for each subject, qualitative comparisons will be made regarding areas of 18F-FDG and 11C-PBR28 uptake, as well as stress, strength, and RPI.
Time Frame: 9-10 months
Population: Because recruitment goals were not met, this computerized numerical method was not completed. We were only able to enroll 2 subjects.
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day.
Description: We were only able to enroll 2 subjects.
Arm/Group | Control Group | Small AAA's | Rapidly Expanding AAA's | AAA's Undergoing Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1 | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03231397/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03231397/ICF_001.pdf